CLINICAL TRIAL: NCT06357104
Title: Detoxification From the Lipid Tract by Cocktail Design
Brief Title: Detoxification From the Lipid Tract
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pachankis, Yang I., M.D. (Individual)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI-CT-0001
Record Dates: First submitted 2024-03-10; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: COVID-19 Vaccine Adverse Reaction
Keywords: sebaceous immunobiology; lipid; depression
MeSH Terms: conditions — Depression | interventions — Deep Brain Stimulation; Sertraline; Clonazepam; Alprazolam; Metoprolol; Adrenergic beta-Antagonists; Olanzapine; Pravastatin; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GABA Cocktail (Experimental)
  Interventions: Device: electroencephalogram biofeedback; Device: electrical brain stimulation; Device: ultra-low frequency transcranial magnetic stimulation; Drug: Sertraline Hydrochloride; Drug: Clonazepam; Drug: Alprazolam; Drug: Metoprolol; Drug: Olanzapine; Drug: Pravastatin Sodium 20 MG; Drug: Sacubitril Valsartan Sodium Hydrate

INTERVENTIONS:
Device: electroencephalogram biofeedback — EB is conducted for 20 minutes per section with two sections per day in the primary efficacy endpoint.
  Other Names: EB
Device: electrical brain stimulation — EBS is conducted for 20 minutes per section per day in the primary efficacy endpoint.
  Other Names: EBS
Device: ultra-low frequency transcranial magnetic stimulation — ULF-TMS is conducted mainly for the left side of the participant's brain for 20 minutes per section per day in the primary efficacy endpoint.
  Other Names: ULF-TMS
Drug: Sertraline Hydrochloride — Sertraline is taken in the morning for 150 mg per day.
  Other Names: SSRI
Drug: Clonazepam — Clonazepam is taken in the morning for 1 mg per day.
Drug: Alprazolam — Alprazolam is introduced near the end of the primary efficacy endpoint for 0.4 mg per night.
Drug: Metoprolol — Metoprolol is introduced at the secondary efficacy endpoint starting with 47.5 mg per night and increase to 95 mg per night.
  Other Names: beta blocker
Drug: Olanzapine — Olanzapine is taken throughout the trial with 7.5 mg per night at first, and increases to 10 mg per night after the cocktail therapy.
Drug: Pravastatin Sodium 20 MG — Pravastatin sodium is introduced in the secondary efficacy endpoint with 20 mg per night.
Drug: Sacubitril Valsartan Sodium Hydrate — Sacubitril valsartan sodium is introduced in the secondary efficacy endpoint with 100 mg per day.
  Other Names: ARNI

SUMMARY:
Apart from electroencephalogram biofeedback and electrical brain stimulation adopted for maintenance treatment, the study utilizes ultra-low frequency transcranial magnetic stimulation (ULF-TMS) for initial γ-aminobutyric acid (GABA) stimulation. The cocktail therapy starts after the primary efficacy endpoint, and concomitant therapy is adopted throughout the study.

DETAILED DESCRIPTION:
It was tested that GABA, in the joint action with topiramate, modulates macrophage activities by modulating cholesterol-metabolism associated molecules. GABA A receptors exhibit highly dynamic trafficking and cell surface mobility and influence on post-endocytic effects. Benzodiazepines (BZDs) exercise the mechanism of action by facilitating the binding of the inhibitory neurotransmitter GABA at various GABA receptors throughout the central nervous system (CNS). Alprazolam, a type of BZD, was tested by Al-Tubuly, Aburawi, Alghzewi, Gorash and Errwami in joint action with water-soluble beta blocker atenolol, in comparison with the non-selective β-adrenoceptor antagonist propranolol on the pharmacological effects on depression. The study hypothesizes that by replacing the water-soluble beta blocker to lipid-soluble one metoprolol, the effect of detoxification from the lipid and sebaceous immunobiological pathways can be achieved by the clathrin-dependent endocytosis process.

Even though partial progress was made in the NCT05839236 trial by statin therapies, the therapeutic effects have not been lasting nor significant. The study develops from the previous protocol for a cocktail therapy by the joint mechanism of actions of alprazolam, metoprolol, and pravastatin sodium for the detoxification process.

ELIGIBILITY:
Inclusion Criteria:

* People who received full doses of COVID-19 vaccines.

Exclusion Criteria:

* Women during pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Changes in Leukocyte and Components' Quantities | 24 days
  All white blood cells are evaluated.
Changes in Leukocyte Components' Ratios | 24 days
  All white blood cells are evaluated.
Quantity Changes in Megakaryocyte-Erythroid Progenitor | 24 days
Changes in Hemoglobin Distribution | 24 days
Changes in Mean Corpuscular Hemoglobin | 24 days
Changes in Hematocrit | 24 days
Changes in Plateletcrit | 24 days
Red cell Distribution Width Coefficient of Variation | 24 days
Changes in Particulate Matter Sizes | 24 days
Changes in Total Lipid Quantities | 24 days
Changes in Apolipoproteina | 24 days
Changes in Lipoprotein (a) | 24 days

SECONDARY OUTCOMES:
Blood Pressure Changes | 24 days
  Recorded systolic and diastolic blood pressures' changes before and after medication each day.
Heart Rate Changes | 24 days
  Heart rate changes before and after medication each day.

CONTACTS AND LOCATIONS:
Locations (1):
- Residential Address, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on Zenodo repository.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Kim H, Nobeyama T, Honda S, Yasuda K, Morone N, Murakami T. Membrane fusogenic high-density lipoprotein nanoparticles. Biochim Biophys Acta Biomembr. 2019 Oct 1;1861(10):183008. doi: 10.1016/j.bbamem.2019.06.007. Epub 2019 Jun 15. PMID 31207206
- [Background] Zhao M, Luo Z, He H, Shen B, Liang J, Zhang J, Ye J, Xu Y, Wang Z, Ye D, Wang M, Wan J. Decreased Low-Density Lipoprotein Cholesterol Level Indicates Poor Prognosis of Severe and Critical COVID-19 Patients: A Retrospective, Single-Center Study. Front Med (Lausanne). 2021 May 26;8:585851. doi: 10.3389/fmed.2021.585851. eCollection 2021. PMID 34124081
- [Background] Glebov OO. Understanding SARS-CoV-2 endocytosis for COVID-19 drug repurposing. FEBS J. 2020 Sep;287(17):3664-3671. doi: 10.1111/febs.15369. Epub 2020 Jun 2. PMID 32428379
- [Background] Pachankis YI. Plausibility Review on Lipoprotein (A) Infection Path of S2 Autoimmune Pathogen. Global Journal of Medical Research. 2023;23(3)(C):5-11.
- [Background] Yang Y, Lian YT, Huang SY, Yang Y, Cheng LX, Liu K. GABA and topiramate inhibit the formation of human macrophage-derived foam cells by modulating cholesterol-metabolism-associated molecules. Cell Physiol Biochem. 2014;33(4):1117-29. doi: 10.1159/000358681. Epub 2014 Apr 9. PMID 24733016
- [Background] Lombardi JP, Kinzlmaier DA, Jacob TC. Visualizing GABA A Receptor Trafficking Dynamics with Fluorogenic Protein Labeling. Curr Protoc Neurosci. 2020 Jun;92(1):e97. doi: 10.1002/cpns.97. PMID 32364672
- [Background] Griffin CE 3rd, Kaye AM, Bueno FR, Kaye AD. Benzodiazepine pharmacology and central nervous system-mediated effects. Ochsner J. 2013 Summer;13(2):214-23. PMID 23789008
- [Background] Al-Tubuly R, Aburawi S, Alghzewi E, Gorash Z, Errwami S. The effect of sympathetic antagonists on the antidepressant action of alprazolam. Libyan J Med. 2008 Jun 1;3(2):78-83. doi: 10.4176/080101. PMID 21499463
- [Background] Hunninghake D, Wallace RB, Reiland S, Barrett-Connor E, Wahl P, Hoover J, Heiss G. Alterations of plasma lipid and lipoprotein levels associated with benzodiazepine use--the LRC Program Prevalence Study. Atherosclerosis. 1981 Oct;40(2):159-65. doi: 10.1016/0021-9150(81)90034-4. PMID 6118165
- [Background] McGrath M, Hoyt H, Pence A, Forman SA, Raines DE. Selective actions of benzodiazepines at the transmembrane anaesthetic binding sites of the GABAA receptor: In vitro and in vivo studies. Br J Pharmacol. 2021 Dec;178(24):4842-4858. doi: 10.1111/bph.15662. Epub 2021 Sep 26. PMID 34386973
- [Background] Mascarenhas FNADP, Silva NF, Menezes-Reis LT, Vieira LG, Hirano LQL, Botelho FV, Ribeiro DL, Zanon RG. Prenatal effects of alprazolam treatment on the immature cerebellum of rats. Int J Dev Neurosci. 2022 Dec;82(8):727-735. doi: 10.1002/jdn.10222. Epub 2022 Aug 5. PMID 35916248
- [Background] Elgarf AA, Siebert DCB, Steudle F, Draxler A, Li G, Huang S, Cook JM, Ernst M, Scholze P. Different Benzodiazepines Bind with Distinct Binding Modes to GABAA Receptors. ACS Chem Biol. 2018 Aug 17;13(8):2033-2039. doi: 10.1021/acschembio.8b00144. Epub 2018 Jul 23. PMID 29767950
- [Background] Pachankis YI. Adrenaline Intolerance in ASD Curing From Autoimmune Pathogens - Sebaceous Immunobiology in Autoimmune Pathogen Research. Biomedical Review: Journal of Basic and Applied Medical Sciences. 2023;10(1):8-14.
- [Background] Kottyan LC, Collier AR, Cao KH, Niese KA, Hedgebeth M, Radu CG, Witte ON, Khurana Hershey GK, Rothenberg ME, Zimmermann N. Eosinophil viability is increased by acidic pH in a cAMP- and GPR65-dependent manner. Blood. 2009 Sep 24;114(13):2774-82. doi: 10.1182/blood-2009-05-220681. Epub 2009 Jul 29. PMID 19641187
- [Background] Petersen OH, Gerasimenko OV, Gerasimenko JV. Endocytic uptake of SARS-CoV-2: the critical roles of pH, Ca2+, and NAADP. Function (Oxf). 2020 Jun 5;1(1):zqaa003. doi: 10.1093/function/zqaa003. eCollection 2020. No abstract available. PMID 38626245
- [Background] Cao Z, Zhao M, Sun H, Hu L, Chen Y, Fan Z. Roles of mitochondria in neutrophils. Front Immunol. 2022 Aug 19;13:934444. doi: 10.3389/fimmu.2022.934444. eCollection 2022. PMID 36081497
- [Background] Fox S, Leitch AE, Duffin R, Haslett C, Rossi AG. Neutrophil apoptosis: relevance to the innate immune response and inflammatory disease. J Innate Immun. 2010;2(3):216-27. doi: 10.1159/000284367. Epub 2010 Feb 11. PMID 20375550
- [Background] Parihar A, Eubank TD, Doseff AI. Monocytes and macrophages regulate immunity through dynamic networks of survival and cell death. J Innate Immun. 2010;2(3):204-15. doi: 10.1159/000296507. Epub 2010 Mar 16. PMID 20375558
- [Background] Salih RQ, Salih GA, Abdulla BA, Ahmed AD, Mohammed HR, Kakamad FH, Salih AM. False-positive HIV in a patient with SARS-CoV-2 infection; a case report. Ann Med Surg (Lond). 2021 Nov;71:103027. doi: 10.1016/j.amsu.2021.103027. Epub 2021 Nov 6. PMID 34777794
- [Background] Robinson MA, Nagurla SR, Noblitt TR, Almaghlouth NK, Al-Rahamneh MM, Cashin LM. Falsely positive fourth generation ADVIA Centaur(R) HIV Antigen/Antibody Combo assay in the presence of autoimmune hepatitis type I (AIH). IDCases. 2020 Jun 25;21:e00886. doi: 10.1016/j.idcr.2020.e00886. eCollection 2020. PMID 32642434
- See also: Benzodiazepines drug profile. European Monitoring Centre for Drugs and Drug Addiction. — https://www.emcdda.europa.eu/publications/drug-profiles/benzodiazepines_en
- See also: Antianxiety Drugs Successfully Treat Autism — http://www.scientificamerican.com/article/antianxiety-drugs-successfully-treat-autism/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT06357104/Prot_ICF_000.pdf